CLINICAL TRIAL: NCT00958464
Title: The Effect of Perthes' Disease on Hip Cartilage
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kishore Mulpuri, Principle Investigator, University of British Columbia
Other Study IDs: H07-00930
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Perthes' Disease
Keywords: MRI; Perthes'disease; hip; cartilage
MeSH Terms: conditions — Legg-Calve-Perthes Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: MRI protocol on 2 separate occasions
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — MRI protocol consists of intravenous injection of 0.4 ml/kg dose of gadopentetate dimeglumine 2- [Gd-DTPA2-] contrast agent (Magnevist, Bayer) 90 minutes prior to imaging.

SUMMARY:
The purpose of this study is to determine whether Perthes' disease has caused detectable hip cartilage damage in young people who have reached the healed stage of the disease.

DETAILED DESCRIPTION:
We will recruit 20 subjects from our healed Perthes' population. We will use dGEMRIC imaging to identify regions of cartilage degeneration in the femur and acetabulum. Both hips will be imaged so that we can use the unaffected side as a control. We will apply dGEMRIC imaging, which allows the composition of cartilage (specifically, the concentration of glycosaminoglycans [GAGs], important structural proteins in the cartilage) to be assessed.

The MRI protocol consists of intravenous injection of 0.4 ml/kg dose of gadopentetate dimeglumine 2- [Gd-DTPA2-] contrast agent (Magnevist, Bayer) 90 minutes prior to imaging. Due to the need to image within a relatively narrow window of time, each hip of each subject must be imaged on separate days. The subject will be asked to walk for 10 minutes after receiving the contrast agent injection to facilitate equilibration of contrast agent into the hip joint.

The scans will be performed at UBC's High Field Imaging Centre on the 3T Phillips Intera scanner. Dr. Wilson has access to this scanner for his research. The scanning protocol is as follows: 3D IR-TFE sequence with TR/TE/Flip of 4.7 ms/1.6 ms/30 o and seven inversion times; 1600, 1200, 800, 400, 200, 300, and 100 ms. In-plane resolution is 0.7 mm with a slice thickness of 3 mm. Total imaging time is approximately 1 hour (at each visit). The T1 calculated image will be obtained using validated, custom written software (IGOR). The resulting image provides a map approximating glycosaminoglycan concentration and, consequently, cartilage degeneration.

The MRI will not be done under sedation. MRIs are performed under sedation at BCCH for children under age seven. Subjects in this study will be between the ages of 7 and 18. The contrast agent, Gd-DTPA2- is routinely used in children in the clinical setting.

Radiographs used for comparison are obtained as part of standard of care follow-up protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have reached the healed stage of unilateral Perthes' disease. -Subjects will be between 7 and 18 years of age.
* Subjects must understand English.

Exclusion Criteria:

* Subjects will be excluded if they have bilateral Perthes' disease or if they have not yet reached the healing stage of the disease.
* Subjects will also be excluded if they do not meet the criteria to have an MRI (e.g., the subject has metal implants, is claustrophobic, has a metallic object in eye or a pacemaker).
* A subject will be excluded if they have any of the precautions for the MR contrast agent, Magnevist, such as pregnancy, breast-feeding, respiratory allergies, asthma, thrombotic syndromes, history of grand mal seizures, impaired renal or hepatic function.

Ages: 17 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Volunteers with healed unilateral Perthes' disease between the ages of 7-18 years
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Whether Perthes' disease has caused detectable hip cartilage damage in young people who have reached the healed stage of the disease. | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Mulpuri, Dr., Principal Investigator — University of British Columbia; David Wilson, Dr., Study Director — University of British Columbia
Locations (1):
- BC Children's Hospital, Department of Orthopaedics, Vancouver, British Columbia, Canada